CLINICAL TRIAL: NCT05985512
Title: A Research on the Typing of Insomnia Disorder Based on Multidimensional Features
Brief Title: Subtyping of Insomnia Disorders Based on Multidimensional Features
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ChengmeiYUAN
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insomnia Disorder (Other): Patients with insomnia disorder
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia is the main therapy for the patients. Medications include sedative-hypnotics and antidepressants with a sedative effect.
  Other Names: Pharmalogical Therapy

SUMMARY:
Based on real world and focusing on patients with chronic sleep disorders, this study conducts a data-driven subtyping research on the clinical symptoms, polysomnography, near-infrared scanning, molecular genetics, and other characteristics of chronic insomnia disorders. It constructs a multimodal therapeutic outcome prediction model, providing a basis for personalized interventions for chronic insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years, regardless of gender;
2. Currently meeting the diagnostic criteria for insomnia disorder according to the Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
3. Pittsburgh Sleep Quality Index (PSQI) total score ≥ 10;
4. Sufficient level of education and comprehension to complete the required examinations and assessments for this study;
5. Voluntarily participating in this research and signing the informed consent form.

Exclusion Criteria:

1. Currently diagnosed with other sleep disorders (sleep-related breathing disorders, periodic limb movement disorder, parasomnias, central disorders of hypersomnolence, circadian rhythm sleep-wake disorders, etc.);
2. Currently diagnosed with organic brain diseases (epilepsy, cerebrovascular disease, etc.) or other organic diseases;
3. Patients with a history of or currently diagnosed with bipolar and related disorders, obsessive-compulsive and related disorders, schizophrenia spectrum and other psychotic disorders, trauma and stressor-related disorders, dissociative disorders, or eating disorders;
4. Women who are pregnant, breastfeeding, or planning to become pregnant during the study period;
5. Insomnia caused by alcohol or substance abuse;
6. High suicide risk, with HAMD-17 suicide factor score > 2;
7. Inability to cooperate with near-infrared examinations and polysomnography due to physical conditions such as head injury, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
polysomnography | the end of the eighth week
  change in total sleep time recorded by polysomnography
PSQI | the end of the 24th, 36th, 48th week
  change in total sleep time according to PSQI scale

CONTACTS AND LOCATIONS:
Overall Officials: Chengmei YUAN, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No